CLINICAL TRIAL: NCT05524948
Title: A Randomized, Single-Blind Clinical Study Assessing the Effects of an Experimental Dentifrice Compared to a Regular Fluoride Dentifrice on Breath Odor When Used Twice Daily for 3 Weeks in a Population With Clinically Diagnosed Gingivitis
Brief Title: A Clinical Study to Examine the Effects of an Experimental Toothpaste Compared to a Regular Fluoride Toothpaste on Breath Odor in a Population With Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300025
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-03

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Dentifrice (Experimental): Participants will be instructed to brush twice daily (for 1 minute, morning and evening) with the experimental dentifrice (0.454% Stannous Fluoride with 0.3% Zinc Chloride) for 3 weeks.
  Interventions: Other: Experimental Dentifrice
- Reference Dentifrice (Active Comparator): Participants will be instructed to brush twice daily (for 1 minute, morning and evening) with the reference dentifrice (Regular Fluoride Dentifrice) for 3 weeks.
  Interventions: Other: Reference Dentifrice

INTERVENTIONS:
Other: Experimental Dentifrice — Dentifrice containing 0.454% stannous fluoride with 0.3% zinc chloride.
  Arms: Experimental Dentifrice
Other: Reference Dentifrice — Standard fluoride dentifrice containing 0.243% sodium fluoride.
  Arms: Reference Dentifrice

SUMMARY:
The purpose of this study is to investigate the efficacy of an experimental dentifrice, containing 0.454 percent (%) stannous fluoride and 0.3% zinc chloride, to reduce oral malodor, compared to a marketed regular fluoride dentifrice after 3 weeks twice daily brushing in a population of clinically diagnosed gingivitis.

DETAILED DESCRIPTION:
This will be a single center, single blind (to the examiners undertaking the oral malodor assessments), randomized (stratified by the participant's sex), controlled, two arm parallel study in volunteers with clinically diagnosed gingivitis and oral malodor. The study will evaluate the clinical efficacy of an experimental dentifrice containing 0.454% stannous fluoride and 0.3% zinc chloride to reduce oral malodor after 3 weeks of twice-daily use compared to a regular reference dentifrice. Sufficient participants will be screened to randomize approximately 106 participants to study treatment (approximately 53 per treatment group) to ensure approximately 100 evaluable participants complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant who is willing and able to comply with scheduled visits, product usage requirements, study procedures and lifestyle restrictions.
* Participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history (for example, a medical condition or medication confirmed to contribute to xerostomia),or upon oral examination, that would impact the participant's safety, wellbeing or the outcomes of the study, if they were to participate in the study, or affect the participant's ability to understand and follow study procedures and requirements.
* Participant with generally good oral health that fulfil all of the following:

  1. Having at least 20 natural (vital) teeth.
  2. Good oral health without lesions in the oral cavity (including the tongue) that could interfere with the study evaluations.
  3. Having clinically diagnosed, plaque-induced gingivitis defined as having 10-30% bleeding sites from the bleeding on probing assessment.
  4. At Screening (Visit 1) and prior to brushing with assigned dentifrice at Baseline (Visit 2) participants must provide 2 samples of mouth air, which must have a mean hydrogen sulfide concentration greater than 150ppb. There must be less than or equal to (<=)500ppb difference between the values measured at screening and baseline (pre-brushing).
  5. At Baseline (Visit 2), prior to brushing with assigned dentifrice participants must provide a breath sample with a mean organoleptic score greater than or equal to (>=)2.

Exclusion Criteria:

* Participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or an employee of the sponsor directly involved in the conduct of the study or a member of their immediate family.
* Participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days of study entry and/or during study participation or who has previously been enrolled in this study.
* Participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A Participant who is pregnant (self-reported) or intending to become pregnant during the study.
* Participant who is breastfeeding.
* Participant who habitually smokes, uses tobacco products or who vapes.
* Participant with known or suspected intolerance or hypersensitivity to the study products or any of their stated ingredients (or closely related compounds).
* Participant who is unwilling or, in the opinion of the investigator or medically qualified designee, unable to comply with the requirements and/or Lifestyle Considerations of the study.
* Participant with a recent history (within the last year) of alcohol or other substance abuse.
* General medical exclusions:

  1. Participant with a medical history that may prevent the Participant from participating in the study until study conclusion.
  2. Participant with, or having recent history of, bronchitis, tonsillitis or sinusitis (within 6 weeks) or any other systemic condition that can cause oral malodor for example, xerostomia, chronic acid reflux, Type 1 diabetes, Crohn's disease, celiac disease or liver/kidney conditions.
  3. Participant with a significant infectious disease, such as hepatitis, COVID-19, flu, respiratory infection, tuberculosis, or any other condition which can be transmitted in saliva or salivary aerosols which, in the opinion of the examiner, could endanger the organoleptic assessors.
  4. Participant with any condition that impacts gum health (for example, Type 2 Diabetes).
* General medication exclusions:

  1. Participant using any antibiotic medication within 14 days prior to screening or at any time during the study.
  2. Participant using chlorhexidine, cetylpyridinium chloride (CPC) or stannous fluoride containing mouthwash or dentifrice within 14 days prior to Visit 2 or between Visit 2 and 3.
  3. Participant taking medications which may impact oral mouth odor (for example, Diazepam, Alprazolam, Lorazepam and so on).
* General oral exclusions:

  1. Participant with orthodontic or prosthetic appliances (fixed or removable), including dental implants.
  2. Participant having had professional dental cleaning (oral prophylaxis) within 3 months prior to the screening visit or at any time during the study.
  3. Participant with signs of active periodontal disease (with probing depth greater than [>]3 millimeter [mm]) or who is receiving or has received treatment for periodontal disease (including surgery) within 12 months of Screening.
  4. Participant who has had oral surgery or tooth extraction within 6 weeks of the screening visit.
  5. Participant who has dental conditions or disease under active dental treatment or requiring immediate treatment.
  6. Participant with tongue or lip piercing.
  7. Participant with Oral Soft Tissue (OST) examination findings at Screening which, in the opinion of the investigator, could interfere with the conduct of the study (for example, stomatitis, open sores, lesions, cavitied caries lesions, redness or swelling).
  8. Participant who does not practice daily oral care.
* Participant with oral malodor which, in the opinion of the investigator, is not expected to respond to treatment with an over-the-counter dentifrice.
* Participant who, in the opinion of the investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at a single center in United States of America (USA).
Pre-assignment Details: A total of 104 participants were screened, enrolled and randomized (52 participants to the experimental dentifrice group and 52 participants to the reference dentifrice group) in the study, of which 101 participants completed the study.
Groups:
- Experimental Dentifrice: In this arm, eligible participants applied a ribbon of experimental dentifrice (0.454 percentage [%] stannous fluoride with 0.3% zinc chloride) to the toothbrush head and brushed their teeth under supervision for one timed minute on Visit 2 (1 to 3 weeks after screening). One hour (+/-5 minutes) post-brushing, participants had their post-brushing assessments and were instructed to brush twice daily (for 1 minute, morning and evening) with experimental dentifrice for the next 3 weeks until their next visit (Visit 3). At Visit 3 (Week 3), participants received the experimental dentifrice and underwent pre-brushing and post-brushing assessments in the same manner as performed at the Visit 2.
- Reference Dentifrice: In this arm, eligible participants applied a ribbon of reference dentifrice (0.243% sodium fluoride) to the toothbrush head and brushed their teeth under supervision for one timed minute on Visit 2 (1 to 3 weeks after screening). One hour (+/-5 minutes) post-brushing, participants had their post-brushing assessments and were instructed to brush twice daily (for 1 minute, morning and evening) with reference dentifrice for the next 3 weeks until their next visit (Visit 3). At Visit 3 (Week 3), participants received the reference dentifrice and underwent pre-brushing and post-brushing assessments in the same manner as performed at the Visit 2.
Period: Overall Study
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Started | 52 | 52
Completed | 50 | 51
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Participant did not receive call or showed up for final visit | 1 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent-To-Treat (mITT) population included all randomized participants who completed at least one use of study product and had at least one post treatment efficacy assessment.
Groups:
- Experimental Dentifrice: In this arm, eligible participants applied a ribbon of experimental dentifrice (0.454% stannous fluoride with 0.3% zinc chloride) to the toothbrush head and brushed their teeth under supervision for one timed minute on Visit 2 (1 to 3 weeks after screening). One hour (+/-5 minutes) post-brushing, participants had their post-brushing assessments and were instructed to brush twice daily (for 1 minute, morning and evening) with experimental dentifrice for the next 3 weeks until their next visit (Visit 3). At Visit 3 (Week 3), participants received the experimental dentifrice and underwent pre-brushing and post-brushing assessments in the same manner as performed at the Visit 2.
- Total: Total of all reporting groups
Arm/Group | Experimental Dentifrice | Reference Dentifrice | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (10.91) | 46.4 (11.17) | 47.4 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 76
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 48 | 51 | 99
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 37 | 43 | 80
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline (Day 0, Pre-Brushing) to Week 3 (Pre-Brushing) in Breath Organoleptic Scores
Description: An organoleptic assessment was used to evaluate the oral odor and defined as a method that measures the strength of target odor and expresses the value in terms of a score with reference to a pre-defined organoleptic scale. The assessors evaluated the oral odor and scored from 0 (lowest score) to 5 (highest score), where 0= No appreciable odor, 1= Barely noticeable odor, 2= Slight but clearly noticeable odor, 3= Moderate odor, 4= Strong odor, 5= Extremely foul odor. Lower score indicates improvement. The change from Baseline was calculated as score at Week 3 (Pre-Brushing) minus score at Baseline (Day 0, Pre-Brushing). Baseline was defined as Day 0 (Pre-Brushing). Analysis was performed using Analysis of Covariance (ANCOVA) method.
Time Frame: Baseline (Day 0, Pre-Brushing) and Week 3 (Pre-Brushing)
Population: mlTT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 50 | 51
Score on a scale | -1.23 (0.146) | 0.07 (0.145)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p < 0.0001, ANCOVA; Analysis was performed using ANCOVA model with study product and gender as a factor and Baseline overall breath organoleptic score as a covariate; Adjusted Mean Difference = -1.30, 95% CI 2-sided [-1.71 to -0.90], Standard Error of Mean 0.206 — Adjusted mean difference was calculated as experimental dentifrice minus reference dentifrice

2. Secondary Outcome: Adjusted Mean Change From Baseline (Day 0, Pre-Brushing) to Week 3 (Pre-Brushing) in Total Volatile Sulfur Compounds (VSCs) Concentration in Breath
Description: The VSCs concentration in breath sample was evaluated using OralChroma Halitosis Measuring instrument. A clean and sterile OralChroma syringe was used to obtain a sample of the mouth air of the participant. The OralChroma is a portable gas chromatograph with a highly sensitive semiconductor gas detector which can determine the concentration of the three main VSCs in breath (hydrogen sulfide, methanethiol and dimethyl sulfide). The concentration values (in parts per billion [ppb]) of hydrogen sulfide, methanethiol and dimethyl sulfide were recorded separately, and the adjusted mean of total VSCs concentration was reported. The change from Baseline was calculated as value at Week 3 (Pre-Brushing) minus value at Baseline (Day 0, Pre-Brushing). Baseline was defined as Day 0 (Pre-Brushing).
Time Frame: Baseline (Day 0, Pre-Brushing) and Week 3 (Pre-Brushing)
Population: mlTT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: Parts per billion
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 50 | 51
Parts per billion | -518.00 (68.469) | 51.64 (67.779)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p < 0.0001, ANCOVA; Analysis was performed using ANCOVA model with study product and gender as a factor and baseline concentration as a covariate; Adjusted Mean Difference = -569.64, 95% CI 2-sided [-763.11 to -376.17], Standard Error of Mean 97.479

3. Secondary Outcome: Adjusted Mean Change From Baseline (Day 0, Pre-Brushing) to Week 3 (Pre-Brushing) in Hydrogen Sulfide, Methanethiol and Dimethyl Sulfide Concentration in Breath
Description: The VSCs concentration in breath sample was evaluated using the OralChroma Halitosis Measuring instrument. A clean and sterile OralChroma syringe was used to obtain a sample of the mouth air of the participant. The OralChroma is a portable gas chromatograph with a highly sensitive semiconductor gas detector which can determine the concentration of the three main VSCs in breath (hydrogen sulfide, methanethiol and dimethyl sulfide). The concentration values (ppb) of hydrogen sulfide, methanethiol and dimethyl sulfide were recorded separately. The change from Baseline was calculated as value at Week 3 (Pre-Brushing) minus value at Baseline (Day 0, Pre-Brushing). Baseline was defined as Day 0 (Pre-Brushing).
Time Frame: Baseline (Day 0, Pre-Brushing) and Week 3 (Pre-Brushing)
Population: mlTT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: Parts per billion
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 50 | 51
Parts per billion
  Hydrogen Sulfide | -348.60 (45.553) | 70.26 (45.093)
  Methanethiol | -118.88 (23.040) | -9.97 (22.810)
  Dimethyl Sulfide | -42.59 (16.234) | -16.42 (16.074)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -418.86, 95% CI 2-sided [-547.56 to -290.15], Standard Error of Mean 64.848 — For Hydrogen Sulfide
Statistical Analysis 2: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p = 0.0012, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -108.90, 95% CI 2-sided [-173.66 to -44.15], Standard Error of Mean 32.626 — For Methanethiol
Statistical Analysis 3: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p = 0.2561, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -26.17, 95% CI 2-sided [-71.64 to 19.29], Standard Error of Mean 22.909 — For Dimethyl Sulfide

4. Secondary Outcome: Adjusted Mean Change From Baseline (Day 0, Pre-Brushing) to Week 3 (1 Hour Post-Brushing) in Total VSC Concentration in Breath
Description: The VSCs concentration in breath sample was evaluated using the OralChroma Halitosis Measuring instrument. A clean and sterile OralChroma syringe was used to obtain a sample of the mouth air of the participant. The OralChroma is a portable gas chromatograph with a highly sensitive semiconductor gas detector which can determine the concentration of the three main VSCs in breath (hydrogen sulfide, methanethiol and dimethyl sulfide). The concentration values (ppb) of hydrogen sulfide, methanethiol and dimethyl sulfide were recorded separately, and the adjusted mean of total VSCs concentration was reported. The change from Baseline was calculated as value at Week 3 (1 Hour Post-Brushing) minus value at Baseline (Day 0, Pre-Brushing). Baseline was defined as Day 0 (Pre-Brushing).
Time Frame: Baseline (Day 0, Pre-Brushing) and Week 3 (1 Hour Post-Brushing)
Population: mlTT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: Parts per billion
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 50 | 51
Parts per billion | -733.17 (66.436) | -11.59 (65.766)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -721.58, 95% CI 2-sided [-909.31 to -533.86], Standard Error of Mean 94.584

5. Secondary Outcome: Adjusted Mean Change From Baseline (Day 0, Pre-Brushing) to Week 3 (1 Hour Post--Brushing) in Hydrogen Sulfide, Methanethiol and Dimethyl Sulfide Concentration in Breath
Description: The VSCs concentration in breath sample was evaluated using the OralChroma Halitosis Measuring instrument. A clean and sterile OralChroma syringe was used to obtain a sample of the mouth air of the participant. The OralChroma is a portable gas chromatograph with a highly sensitive semiconductor gas detector which can determine the concentration of the three main VSCs in breath (hydrogen sulfide, methanethiol and dimethyl sulfide). The concentration values (ppb) of hydrogen sulfide, methanethiol and dimethyl sulfide were recorded separately. The change from Baseline was calculated as value at Week 3 (1 Hour Post-Brushing) minus value at Baseline (Day 0, Pre-Brushing). Baseline was defined as Day 0 (Pre-Brushing).
Time Frame: Baseline (Day 0, Pre-Brushing) and Week 3 (1 Hour Post-Brushing)
Population: mlTT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: Parts per billion
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 50 | 51
Parts per billion
  Hydrogen Sulfide | -507.84 (47.830) | 60.05 (47.348)
  Methanethiol | -176.69 (17.351) | -71.30 (17.178)
  Dimethyl Sulfide | -43.45 (18.568) | -5.42 (18.384)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -567.89, 95% CI 2-sided [-703.03 to -432.75], Standard Error of Mean 68.090 — For Hydrogen Sulfide
Statistical Analysis 2: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -105.39, 95% CI 2-sided [-154.15 to -56.62], Standard Error of Mean 24.570 — For Methanethiol
Statistical Analysis 3: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p = 0.1498, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -38.04, 95% CI 2-sided [-90.04 to 13.97], Standard Error of Mean 26.201 — For Dimethyl Sulfide

6. Secondary Outcome: Adjusted Mean Change From Baseline (Day 0, Pre-Brushing) to Week 3 (1 Hour Post-Brushing) in Breath Organoleptic Scores
Description: An organoleptic assessment was used to evaluate the oral odor and defined as a method that measures the strength of target odor and expresses the value in terms of a score with reference to a pre-defined organoleptic scale. The assessors evaluated the oral odor and scored from 0 (lowest score) to 5 (highest score), where 0= No appreciable odor, 1= Barely noticeable odor, 2= Slight but clearly noticeable odor, 3= Moderate odor, 4= Strong odor, 5= Extremely foul odor. Lower score indicates improvement. The change from Baseline was calculated as score at Week 3 (1 Hour Post-Brushing) minus score at Baseline (Day 0, Pre-Brushing). Baseline was defined as Day 0 (Pre-Brushing).
Time Frame: Baseline (Day 0, Pre-Brushing) and Week 3 (1 Hour Post-Brushing)
Population: mlTT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 50 | 51
Score on a scale | -2.55 (0.145) | -0.38 (0.143)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Mean Difference = -2.17, 95% CI 2-sided [-2.58 to -1.77], Standard Error of Mean 0.204 — Adjusted mean difference was calculated as experimental dentifrice minus reference dentifrice

7. Secondary Outcome: Adjusted Mean Change From Baseline (Day 0, Pre-Brushing) to Day 0 (1 Hour Post-Brushing) in Total VSC Concentration in Breath
Description: The VSCs concentration in breath sample was evaluated using the OralChroma Halitosis Measuring instrument. A clean and sterile OralChroma syringe was used to obtain a sample of the mouth air of the participant. The OralChroma is a portable gas chromatograph with a highly sensitive semiconductor gas detector which can determine the concentration of the three main VSCs in breath (hydrogen sulfide, methanethiol and dimethyl sulfide). The concentration values (ppb) of hydrogen sulfide, methanethiol and dimethyl sulfide were recorded separately, and the adjusted mean of total VSCs concentration was reported. The change from Baseline was calculated as value at Day 0 (1 Hour Post-Brushing) minus value at Baseline (Day 0, Pre-Brushing). Baseline was defined as Day 0 (Pre-Brushing).
Time Frame: Baseline (Day 0, Pre-Brushing) and Day 0 (1 Hour Post-Brushing)
Population: mITT population.
Measure: Mean (Standard Error); unit: Parts per billion
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 52 | 52
Parts per billion | -434.60 (67.213) | -37.64 (67.213)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -396.96, 95% CI 2-sided [-586.51 to -207.41], Standard Error of Mean 95.541

8. Secondary Outcome: Adjusted Mean Change From Baseline (Day 0, Pre-Brushing) to Day 0 (1 Hour Post-Brushing) in Hydrogen Sulfide, Methanethiol and Dimethyl Sulfide Concentration in Breath
Description: The VSCs concentration in breath sample was evaluated using the OralChroma Halitosis Measuring instrument. A clean and sterile OralChroma syringe was used to obtain a sample of the mouth air of the participant. The OralChroma is a portable gas chromatograph with a highly sensitive semiconductor gas detector which can determine the concentration of the three main VSCs in breath (hydrogen sulfide, methanethiol and dimethyl sulfide). The concentration values (ppb) of hydrogen sulfide, methanethiol and dimethyl sulfide were recorded separately. The change from Baseline was calculated as value at Day 0 (1 Hour Post-Brushing) minus value at Baseline (Day 0, Pre-Brushing). Baseline was defined as Day 0 (Pre-Brushing).
Time Frame: Baseline (Day 0, Pre-Brushing) and Day 0 (1 Hour Post-Brushing)
Population: mITT population.
Measure: Mean (Standard Error); unit: Parts per billion
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 52 | 52
Parts per billion
  Hydrogen Sulfide | -324.07 (50.984) | 17.30 (50.984)
  Methanethiol | -137.61 (14.737) | -63.46 (14.737)
  Dimethyl Sulfide | 31.79 (18.313) | 3.81 (18.313)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -341.37, 95% CI 2-sided [-485.10 to -197.64], Standard Error of Mean 72.446 — For Hydrogen Sulfide
Statistical Analysis 2: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p = 0.0006, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -74.15, 95% CI 2-sided [-115.62 to -32.68], Standard Error of Mean 20.905 — For Methanethiol
Statistical Analysis 3: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p = 0.2834, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = 27.98, 95% CI 2-sided [-23.49 to 79.45], Standard Error of Mean 25.942 — For Dimethyl Sulfide

9. Secondary Outcome: Adjusted Mean Change From Baseline (Day 0, Pre-Brushing) to Day 0 (1 Hour Post-Brushing) in Breath Organoleptic Scores
Description: An organoleptic assessment was used to evaluate the oral odor and defined as a method that measures the strength of target odor and expresses the value in terms of a score with reference to a pre-defined organoleptic scale. The assessors evaluated the oral odor and scored from 0 (lowest score) to 5 (highest score), where 0= No appreciable odor, 1= Barely noticeable odor, 2= Slight but clearly noticeable odor, 3= Moderate odor, 4= Strong odor, 5= Extremely foul odor. Lower score indicates improvement. The change from Baseline was calculated as score at Day 0 (1 Hour Post-Brushing) minus score at Baseline (Day 0, Pre-Brushing). Baseline was defined as Day 0 (Pre-Brushing).
Time Frame: Baseline (Day 0, Pre-Brushing) and Day 0 (1 Hour Post-Brushing)
Population: mITT population.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 52 | 52
Score on a scale | -2.11 (0.098) | -0.56 (0.098)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Mean Difference = -1.55, 95% CI 2-sided [-1.83 to -1.28], Standard Error of Mean 0.138 — Adjusted mean difference was calculated as the experimental dentifrice minus the reference dentifrice

10. Secondary Outcome: Adjusted Mean Change From Baseline (Week 3, Pre-Brushing) to Week 3 (1 Hour Post-Brushing) in Total VSC Concentration in Breath
Description: The VSCs concentration in breath sample was evaluated using the OralChroma Halitosis Measuring instrument. A clean and sterile OralChroma syringe was used to obtain a sample of the mouth air of the participant. The OralChroma is a portable gas chromatograph with a highly sensitive semiconductor gas detector which can determine the concentration of the three main VSCs in breath (hydrogen sulfide, methanethiol and dimethyl sulfide). The concentration values (ppb) of hydrogen sulfide, methanethiol and dimethyl sulfide were recorded separately, and the adjusted mean of total VSCs concentration was reported. The change from Baseline was calculated as value at Week 3 (1 Hour Post-Brushing) minus value at Baseline (Week 3, Pre-Brushing). Baseline was defined as Week 3 (Pre-Brushing).
Time Frame: Baseline (Week 3, Pre-Brushing) and Week 3 (1 Hour Post-Brushing)
Population: mlTT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: Parts per billion
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 50 | 51
Parts per billion | -301.42 (47.053) | 21.33 (46.567)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -322.75, 95% CI 2-sided [-457.27 to -188.23], Standard Error of Mean 67.778

11. Secondary Outcome: Adjusted Mean Change From Baseline (Week 3, Pre-Brushing) to Week 3 (1 Hour Post-Brushing) in Hydrogen Sulfide, Methanethiol and Dimethyl Sulfide Concentration in Breath
Description: The VSCs concentration in breath sample was evaluated using the OralChroma Halitosis Measuring instrument. A clean and sterile OralChroma syringe was used to obtain a sample of the mouth air of the participant. The OralChroma is a portable gas chromatograph with a highly sensitive semiconductor gas detector which can determine the concentration of the three main VSCs in breath (hydrogen sulfide, methanethiol and dimethyl sulfide). The concentration values (ppb) of hydrogen sulfide, methanethiol and dimethyl sulfide were recorded separately. The change from Baseline was calculated as value at Week 3 (1 Hour Post-Brushing) minus value at Baseline (Week 3, Pre-Brushing). Baseline was defined as Week 3 (Pre-Brushing).
Time Frame: Baseline (Week 3, Pre-Brushing) and Week 3 (1 Hour Post-Brushing)
Population: mlTT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: Parts per billion
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 50 | 51
Parts per billion
  Hydrogen Sulfide | -210.39 (29.608) | 39.94 (29.300)
  Methanethiol | -82.58 (16.472) | -37.05 (16.307)
  Dimethyl Sulfide | -11.38 (18.470) | 21.31 (18.287)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -250.33, 95% CI 2-sided [-335.35 to -165.30], Standard Error of Mean 42.838 — For Hydrogen Sulfide
Statistical Analysis 2: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p = 0.0550, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -45.53, 95% CI 2-sided [-92.05 to 0.99], Standard Error of Mean 23.439 — For Methanethiol
Statistical Analysis 3: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p = 0.2124, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -32.68, 95% CI 2-sided [-84.36 to 18.99], Standard Error of Mean 26.036 — For Dimethyl Sulfide

12. Secondary Outcome: Adjusted Mean Change From Baseline (Week 3, Pre-Brushing) to Week 3 (1 Hour Post-Brushing) in Breath Organoleptic Scores
Description: An organoleptic assessment was used to evaluate the oral odor and defined as a method that measures the strength of target odor and expresses the value in terms of a score with reference to a pre-defined organoleptic scale. The assessors evaluated the oral odor and scored from 0 (lowest score) to 5 (highest score), where 0= No appreciable odor, 1= Barely noticeable odor, 2= Slight but clearly noticeable odor, 3= Moderate odor, 4= Strong odor, 5= Extremely foul odor. Lower score indicates improvement. The change from Baseline was calculated as score at Week 3 (1 Hour Post-Brushing) minus score at (Week 3, Pre-Brushing). Baseline was defined as Week 3 (Pre-Brushing).
Time Frame: Baseline (Week 3, Pre-Brushing) and Week 3 (1 Hour Post-Brushing)
Population: mlTT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Experimental Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 50 | 51
Score on a scale | -1.49 (0.108) | -0.29 (0.107)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Reference Dentifrice; Test type: Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Mean Difference = -1.20, 95% CI 2-sided [-1.52 to -0.87], Standard Error of Mean 0.164 — Adjusted mean difference was calculated as experimental dentifrice minus reference dentifrice

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious Adverse Events (SAEs), Non-SAEs and Medical Device incidents were collected immediately after signing of informed consent until 5 days following last administration of the study product (Visit 3, Week 3) (Collected up to 35 days)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). A SAE is a particular category of an adverse event where the adverse outcome is serious.
Arm/Group | Experimental Dentifrice | Reference Dentifrice
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-09-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT05524948/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT05524948/SAP_001.pdf